CLINICAL TRIAL: NCT03470805
Title: Phase-II Study of Olaparib as Maintenance Therapy After Response to Trabectedin-pegylated Liposomal Doxorubicin in Recurrent Ovarian Carcinoma
Brief Title: Olaparib After Response to Trabectedin-pegylated Liposomal Doxorubicin in Recurrent Ovarian Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: AstraZeneca (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLATRA; 2017-003183-13 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-20 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: Olaparib as maintenance therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): Olaparib orally twice daily at 150 mgs bid continually
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib will be dispensed to patients on Day 1 and every 28 days thereafter until disease progression, unacceptable toxicity, withdraws from the study or closure of the study

SUMMARY:
Epithelial ovarian cancer harbours 20% Breast Cancer gene (BRCA)1/2 mutations independently of family history. Poly ADP ribose polymerase (PARP) inhibitors (PARPi) have shown clinical activity among patients with homologous recombination deficiency (HRD) and specifically among BRCA1/2 mutation carriers.

The European Medicines Agency (EMA) approved the use of olaparib as maintenance therapy "as monotherapy for the maintenance treatment of adult patients with platinum sensitive relapsed BRCA mutated (germline and/or somatic) high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete response or partial response) to platinum-based chemotherapy".

Trabectedin and Pegylated liposomal doxorubicin (PLD) have shown relevant activity in relapsed epithelial ovarian cancer. In the relapse with Treatment-free interval of last platinum (TFIp) between 6 and 12 months this efficacy translated into an increase in Overall survival (OS) and Progression free survival (PFS).

There is an increase of hypersensitivity reactions (HSR) among platinum sensitive patients, that reaches 44% in third line and does not always allow for platinum use despite desensitization protocols. In relapse with TFIp between 6-12 months the use of Trabectedin+PLD is accepted in guidelines and consensus.

Following clinical BRCAness criteria a group of patients that harbours up to 50% of BRCA1/2 mutations can be selected. Olaparib has been licensed according to EMA for maintenance in BRCA mutated patients after response to platinum following Study 19 phase II trial and further confirmed with phase III SOLO-2 data. However there is no evidence of the benefit of adding olaparib after Trabectedin+PLD response among BRCA1/2 carriers.

The combination of Trabectedin+PLD, as well as both single drugs, have shown higher activity among BRCA1/2 carriers.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Female aged ≥18 years.
3. Patients with high-grade serous or endometrioid ovarian carcinoma.
4. Treatment-free interval of last platinum (TFIp) higher than 6 months.
5. BRCA1/2 germline or somatic deleterious mutation.
6. Patient must have received two or more previous chemotherapy (CT) regimens, including first line platinum based CT and last trabectedin + PLD. There is no limit of previous number of CT lines.
7. Last CT prior to the inclusion in the trial must be trabectedin + PLD. Patients must have received at least 4 cycles of treatment, and have reached a partial or complete response, assessed by RECIST 1.1 criteria and no evidence of a rising CA 125, following the chemotherapy course.
8. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
   * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
10. Life expectancy ≥ 16 weeks.
11. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
13. Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer must be available for central testing if sBRCA analysis is not available at study site. If there is not written confirmation of the availability of an archived tumour sample or gBRCA test performed prior to enrolment the patient is not eligible for the study.

For inclusion in i) the optional exploratory genetic research and ii) the optional biomarker research, patients must fulfil the following criteria:

* Provision of informed consent for genetic research
* Provision of informed consent for biomarker research

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site).
2. Any previous treatment with PARP inhibitor.
3. Rising CA125 after chemotherapy is finished until inclusion. Pre-treatment CA-125 measurements must meet criterion specified below:

   * If the first value is within upper limit of normal (ULN) the patient is eligible to be randomised and a second sample is not required.
   * If the first value is greater than ULN a second assessment must be performed at least 7 days after the first. If the second assessment is ≥ 15% more than the first, the patient is not eligible.
4. Other malignancy within the last 3 years except: adequately treated non-melanoma skin cancer, curatively treated cervical carcinoma in situ, breast carcinoma in situ, and grade 1 endometrial carcinoma in stage 1.
5. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
6. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
7. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St Johns Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
8. Persistent toxicities (> Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
9. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of these diseases.
10. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
11. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
12. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
13. Patients considered a poor medical condition due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
14. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Breast feeding women.
16. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
17. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
18. Patients with known active hepatitis (i.e. Hepatitis B or C).
19. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
20. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 9 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 24 months
  Time from date of first olaparib dose until the date of objective radiological disease progression according to modified RECIST 1.1 or death (by any cause in the absence of progression).

SECONDARY OUTCOMES:
Time to First Subsequent Treatment (TFST) | Up to 24 months
  Time from date of first olaparib dose (treatment initiation) to date of first subsequent treatment commencement or death due to any cause if this occurs before commencement of first subsequent treatment
Time to Second Subsequent Treatment (TSST) | Up to 24 months
  Time from date of first olaparib dose (treatment initiation) to date of second subsequent treatment commencement or death due to any cause if this occurs before commencement of second subsequent treatment.
Progression free survival 2 (PFS2) | Up to 24 months
  Interval from the first olaparib dose (treatment initiation) to the earliest of the progression events subsequent to that used for the primary variable PFS, or death
Incidence of Treatment Adverse Events | Up to 24 months
  Number of Adverse Events per patient

OTHER OUTCOMES:
Predictive biomarkers of long PFS | Up to 24 months
  Gene Mutations

CONTACTS AND LOCATIONS:
Overall Officials: Andres Redondo, MD, Principal Investigator — Hospital La Paz; Ignacio Romero, MD, Principal Investigator — Fundacion Instituto Valenciano de Oncologia
Locations (16):
- Spain (16):
  - ICO Badalona, Badalona
  - H Reina Sofía Cordoba, Córdoba
  - Hospital de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario La Paz, Madrid
  - Fundación Jimenez Diaz, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clinico Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen Macarena, Seville
  - Instituto Valenciano de Oncología, Valencia